CLINICAL TRIAL: NCT07267234
Title: PRaG-1 Plus PRaG Therapy in Advanced Solid Tumors: A Prospective Clinical Trial (PRaG 10.0)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JD-LK2025017-IR01
Record Dates: First submitted 2025-11-24; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Solid Cancer; Lymphopenia; Radiotherapy; Immune Checkpoint Inhibitor
MeSH Terms: conditions — Lymphopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment (Experimental)
  Interventions: Drug: PD -1/PD-L1 monoclonal antibody

INTERVENTIONS:
Drug: PD -1/PD-L1 monoclonal antibody — PRaG-1 Cordycepin Tablets+ Radiotherapy+ GM-CSF+ PD-1/PD-L1 inhibitors

SUMMARY:
The goal of this clinical trial is to learn if a combination treatment using PRaG-1 Cordycepin Tablets with radiation therapy, immune-boosting injections, and immunotherapy drugs can help patients with advanced solid tumors. It will also assess safety. The main questions it aims to answer are:

Does this treatment improve immune function and slow tumor growth? What side effects or risks occur during treatment?

Participants will:

Take PRaG-1 Cordycepin Tablets (a natural compound derived from Cordyceps fungus) orally: higher dose for 7 days before radiation, then lower daily dose for 2 weeks Receive targeted radiation therapy to the tumor area (5-12 Gy total in 2-3 sessions) Get daily immune-boosting injections (GM-CSF) for 7 days starting with radiation Receive immunotherapy drugs (PD-1/PD-L1 inhibitors) within one week after radiation Have blood drawn and small tumor tissue samples taken before and after the first two treatment cycles for immune analysis All participants will receive this combination treatment; there is no placebo or alternative treatment group in this study.

DETAILED DESCRIPTION:
1. This clinical study utilizes PRaG-1 Cordycepin Tablets (oral administration) to modulate immune cell and cytokine profiles. Lymphocyte subset analysis is performed before and after treatment to quantify immune function changes.
2. Treatment phases:

   Cordycepin: PRaG-1 Cordycepin Tablets (manufactured by Life Origin Biotechnology Co., Ltd., affiliated with the National Bioengineering Engineering Technology Center, Nanjing Tech University) contain 200 mg cordycepin per tablet and hold National Food Production License No. SC11332019200201.

   Loading dose: Initiated 1 week prior to radiotherapy, administered as 2 tablets once daily after meals with water for 7 consecutive days.

   Maintenance dose: Following loading dose completion, 1 tablet once daily after meals with water is continued starting with radiotherapy for 2 weeks per cycle (every 3 weeks). Efficacy is assessed at each cycle.

   Biospecimen collection: 5 mL blood and 2 g tumor biopsy tissue are obtained before and after the first two treatment cycles for immune function analysis (including bulk RNA sequencing, single-cell sequencing, TCR sequencing, proteomic analysis, metabolomic analysis, gut microbiome analysis, and urinary extracellular vesicle analysis).

   Treatment discontinuation criteria: Confirmed disease progression, intolerable toxicity, withdrawal of informed consent, death, or other protocol-specified criteria.

   Radiotherapy: Begins on Day 1 of the treatment cycle; 5-12 Gy total dose delivered in 2-3 fractions per lesion, once daily.

   GM-CSF: 200 μg subcutaneously daily starting on radiotherapy day, continued for 7 days.

   Immunotherapy: PD-1/PD-L1 inhibitors initiated within one week post-radiotherapy.
3. Maintenance phases:

Stage A: ≥2 cycles of cordycepin combined with radiotherapy, PD-1/PD-L1 inhibitors, and GM-CSF.

Stage B: Maintenance therapy with PD-1/PD-L1 inhibitors, GM-CSF, and cordycepin for ≥6 months.

Stage C: Continued PD-1/PD-L1 inhibitor monotherapy until disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Histologically confirmed treatment-naïve or relapsed/metastatic advanced solid malignancies with no standard treatment option per current clinical guidelines or intolerance to standard therapy; measurable metastatic lesions ≥1 cm (by RECIST criteria); absolute lymphocyte count (ALC) below lower limit of normal (LLN).
3. No history of congestive heart failure, unstable angina, or unstable cardiac arrhythmias within the past 6 months.
4. ECOG performance status 0-3; estimated life expectancy ≥3 months.
5. No history of significant hematologic, cardiac, pulmonary, hepatic, or renal dysfunction.
6. Baseline AST ≤3×ULN and ALT ≤3×ULN (≤5×ULN for hepatocellular carcinoma or liver metastases); creatinine ≤3×ULN.
7. Capacity to comprehend study procedures and voluntarily provide written informed consent.

Exclusion Criteria:

1. History of other malignancies within the past 5 years, except for adequately treated non-melanoma skin cancer or cervical carcinoma in situ.
2. Uncontrolled epilepsy, central nervous system disorders, or psychiatric disorders that, in the investigator's judgment, may interfere with informed consent or treatment adherence.
3. Clinically significant active cardiac disease, including symptomatic coronary artery disease, NYHA Class II or higher congestive heart failure, severe arrhythmias requiring pharmacological intervention, or myocardial infarction within the past 12 months.
4. History of solid organ transplant requiring ongoing immunosuppressive therapy.
5. Known significant active infection, or significant hematologic, renal, metabolic, gastrointestinal, or endocrine dysfunction, or other serious uncontrolled comorbidities as determined by the investigator.
6. Allergy to any component of the study drug(s).
7. History of immunodeficiency, including HIV infection, acquired or congenital immunodeficiency disorders, solid organ transplant, or chronic immunosuppressive therapy for immune-related conditions.
8. Active or latent tuberculosis infection confirmed by positive T-SPOT.TB test or chest X-ray findings suggestive of tuberculosis.
9. Any other condition that, in the investigator's clinical judgment, may compromise study participation or safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate #ORR# | 36 months
  Objective Response Rate was defined as the percentage of participants with a complete response (CR) or partial response (PR).

SECONDARY OUTCOMES:
Disease control rate (DCR) | 36 months
  DCR was defined as the percentage of participants with a complete response (CR), partial response (PR), or stable disease (SD).
Progression-free Survival (PFS) | 36 months
  PFS was defined as the time from the first administration of study treatment to the first occurrence of disease progression as determined by investigator using RECIST v1.1 or death from any cause, whichever comes first.
Adverse event | 36 months
  rate of adverse events